CLINICAL TRIAL: NCT04816292
Title: A Comparison of the Resection Rate for Hot and Cold Snare Polypectomy of Colorectal Polyps (10-15 Mm) - a Randomized Controlled Trial (COLDSNAP-2)
Brief Title: A Comparison of the Resection Rate for Hot and Cold Snare Polypectomy of Colorectal Polyps (10-15 Mm)
Acronym: COLDSNAP-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Veit Phillip, Departement for Interdisciplinary Endoscopy, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-90-S-P
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Adenomatous Polyps
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hot Snare Polypectomy (Active Comparator): If an eligible polyp 10-15 mm (as compared by the size of the snare) is found, according to the randomized group, HSP is performed for the removal of all eligible polyps in this patient. After polypectomy, the resection site is washed thoroughly with saline water. After the endoscopist carefully examines the resection site for residual adenomatous tissue, eventually another resection with the same method is indicated. Afterwards 4 biopsies (polyps 10-15mm) are performed from the resection margin to reveal presence or absence of residual neoplastic tissue.
  Interventions: Procedure: Active Comparator: Hot Snare Polypectomy
- Cold Snare Polypectomy (Experimental): If an eligible polyp 10-15 mm (as compared by the size of the snare) is found, according to the randomized group, CSP is performed for the removal of all eligible polyps in this patient. After polypectomy, the resection site is washed thoroughly with saline water. After the endoscopist carefully examines the resection site for residual adenomatous tissue, eventually another resection with the same method is indicated. Afterwards 4 biopsies (polyps 10-15mm) are performed from the resection margin to reveal presence or absence of residual neoplastic tissue.
  Interventions: Procedure: Experimental: Cold Snare Polypectomy

INTERVENTIONS:
Procedure: Active Comparator: Hot Snare Polypectomy — Hot Snare Polypectomy with the use of electrocautery for the resection of polyps.
  Arms: Hot Snare Polypectomy
Procedure: Experimental: Cold Snare Polypectomy — Cold Snare Polypectomy without the use of electrocautery for the resection of polyps.
  Arms: Cold Snare Polypectomy

SUMMARY:
Colorectal cancer (CRC) has become the third most common malignant tumor and is the second leading cause of cancer related deaths worldwide. Adenomatous polyps of the colon are possible precursor lesions for CRC. Screening for CRC has been shown effective in preventing CRC and related deaths, especially colonoscopy and resection of adenomatous polyps. Currently, for intermediate sized polyps 5 - 19 mm hot snare polypectomy (HSP) with the use of electrocautery is conventionally used, causing relevant adverse events including haemorrhage and postpolypectomy coagulation syndrome, but is safe regarding complete resection of the polyp due to burning effect on residual tissue. On the other hand, cold snare polypectomy (CSP) has grown popularity. Absence of electrocautery makes it technically easier and most important reduces adverse events. CSP is recommended as the preferred technique for polyps <5 mm by the European Society of Gastrointestinal Endoscopy (ESGE) guidelines. In literature, there is one multicenter trial from Japan recommending CSP for polyps 4-9 mm (average polyp size 5,4 mm) and only a few case studies for polyps 10-15 mm with inconsistent results, especially regarding the complete resection and pathological evaluation of the specimen.

In this randomized controlled trial, the investigators want to compare the complete resection rates of small and intermediate sized colorectal polyps 10-15 mm with CSP and HSP.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colonoscopy
* at least 1 adenomatous polyp 10-15 mm
* provided written informed consent

Exclusion Criteria:

* American Society of Anaesthesiologists class IV or higher
* florid inflammatory bowel disease
* emergency indication for colonoscopy
* haemorrhagic diathesis
* continued dual antiplatelet therapy
* continued anticoagulant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | 6 months
  The histological complete resection rate, determined by pathologically negative margins of the specimen and no residual adenomatous material obtained from two/four biopsies of the resection site.

SECONDARY OUTCOMES:
En-bloc resection rate | During procedure
  Number of additional resections (snare/forceps) needed.
Rate of immediate bleeding with necessity of haemostasis | During procedure
  Immediate bleeding: Bleeding >30 seconds after snaring.
Rate of impossible resection by CSP | During procedure
  An impossible resection by CSP needs electrocautery for successful resection.
Time required for resection | During procedure
  Time required for resection is the time between the insertion of the snare into working channel to the end of polyp resection. In the HSP group, it is defined as the start of submucosal injection until the end of polyp resection.
Rate of procedure-related adverse events. | 6 months
  Delayed bleeding, defined as haemorrhage after colonoscopy with the necessity of endoscopic haemostasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik und Poliklinik für Innere Medizin II, Klinikum rechts der Isar, Technische Universität München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No